CLINICAL TRIAL: NCT05562661
Title: A Randomized, Controlled Clinical Trial of M89PF in Rosacea Associated With Erythema and Sensitive Skin
Brief Title: M89PF in Rosacea Associated With Erythema and Sensitive Skin
Status: Completed | Type: Observational
Sponsor: Cosmetique Active International (Industry)
Responsible Party: Sponsor
Other Study IDs: M89PF splitface
Record Dates: First submitted 2022-09-25; First posted 2022-10-03 (Actual); Last update posted 2022-10-03 (Actual); Status verified 2022-09

CONDITIONS: Rosacea
Keywords: rosacea; skin barrier; exposome; M89PF; splitface; sensitive skin
MeSH Terms: conditions — Rosacea

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- M89PF/standard skin care: use of M89PF on one side of the face standard skin care products on the other side of the face

SUMMARY:
Rosacea is a common facial dermatosis, with flares induced by exposome factors. M89PF containing Vichy mineralizing water, probiotic fractions, hyaluronic acid, niacinamide and tocopherol repairs the skin barrier and reinforces skin defences against exposome factors.

This study assessed the benefit of M89PF in patients with rosacea associated with erythema and sensitive skin during the Covid-19 pandemic with use of protective face masks.

DETAILED DESCRIPTION:
M89PF was compared to usual skin care in a randomized, split-face study, for 30 days in subjects with rosacea associated with erythema and sensitive skin. Clinical evaluations included erythema, desquamation, skin tightness, dryness, burning sensation, itching, stinging, stinging test, and local tolerability. Instrument evaluations included erythema, skin hydration and TEWL. Subject satisfaction was also assessed.

ELIGIBILITY:
Inclusion Criteria:

Adult subjects with rosacea associated with erythema and less than 3 papules or pustules and having sensitive skin (positive 15% lactic acid sting test)

Exclusion Criteria:

None

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult subjects with rosacea associated with erythema and less than 3 papules or pustules and having sensitive skin (positive 15% lactic acid sting test)
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2021-01-02 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
erythema | Day 0
  assessment using a chromameter
erythema | Day 15
  assessment using a chromameter
erythema | Day 30
  assessment using a chromameter
skin hydration | Day 0
  using a corneometer
skin hydration | Day 15
  using a corneometer
skin hydration | Day 30
  using a corneometer
transepidermal water loss | Day 0
  tewameter
transepidermal water loss | Day 15
  tewameter
transepidermal water loss | Day 30
  tewameter

SECONDARY OUTCOMES:
clinical symptoms (skin tightness, dryness, burning sensation, itching and stinging) | Day 0
  VAS 0=none to 10=very severe
clinical symptoms (skin tightness, dryness, burning sensation, itching and stinging) | Day 15
  VAS 0=none to 10=very severe
clinical symptoms (skin tightness, dryness, burning sensation, itching and stinging) | Day 30
  VAS 0=none to 10=very severe
skin sensitivity | Day 0
  lactic acid skin stinging test
skin sensitivity | Day 15
  lactic acid skin stinging test
skin sensitivity | Day 30
  lactic acid skin stinging test
Demodex density | Day 0
  SSSB method
Demodex density | Day 30
  SSSB method
local tolerability | Day 15
  AE questioning
local tolerability | Day 30
  AE questioning
subject satisfaction | Day 15
  questionnaire on a scale from 0= very unsatisfied to 5 very satisfied
subject satisfaction | Day 30
  questionnaire on a scale from 0= very unsatisfied to 5 very satisfied

CONTACTS AND LOCATIONS:
Overall Officials: Delphine Kerob, MD, Study Director — Laboratoires Vichy, Levallois-Perret France
Locations (1):
- ISPE, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Berardesca E, Bonfigli A, Cartigliani C, Kerob D, Tan J. A Randomized, Controlled Clinical Trial of a Dermocosmetic Containing Vichy Volcanic Mineralizing Water and Probiotic Fractions in Subjects with Rosacea Associated with Erythema and Sensitive Skin and Wearing Protective Masks. Clin Cosmet Investig Dermatol. 2023 Jan 11;16:71-77. doi: 10.2147/CCID.S391893. eCollection 2023. PMID 36660190